CLINICAL TRIAL: NCT04883710
Title: The World Federation of Hemophilia Gene Therapy Registry
Acronym: WFH GTR
Status: Not yet recruiting | Type: Observational
Sponsor: World Federation of Hemophilia (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-001
Record Dates: First submitted 2020-02-20; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia
Keywords: Gene therapy
MeSH Terms: conditions — Hemophilia A | interventions — Genetic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gene therapy — This is a prospective patient registry.

SUMMARY:
The aim of the WFH GTR is to provide a database in which long-term data on PWH who receive gene therapy from around the world, will be collected and housed.

DETAILED DESCRIPTION:
The first gene therapy product for hemophilia is expected to receive marketing authorization in 2020, with several others following closely behind. With these new therapies hitting the market in the near future, it is incumbent on us as a community to ensure that we have measures in place to allow monitoring of expected, unexpected and unknown safety issues, as well as duration of efficacy, over the long term. Low incidence adverse events require monitoring of a large number of patients, over a long period of time, necessitating a global initiative.

To fill this need, the World Federation of Hemophilia (WFH), under the guidance of a multi-stakeholder steering committee, is developing and implementation the WFH Gene Therapy Registry (GTR). The aim of the WFH GTR is to provide a database in which long-term data on PWH who receive gene therapy from around the world, will be collected and housed.

The WFH GTR steering committee is made up of hematologists, clinical trialists, methodologists, epidemiologists, manufacturers and patient advocates. All stakeholders have a role in ensuring the success of this important initiative.

The WFH GTR will collect a core set of demographic, safety and efficacy data, on all patients with hemophilia, who receive a gene therapy product via a clinical trial or post-marketing, from anywhere in the world. The core data set is currently in development; and the global implementation plan is being finalized. A database provider will be selected in Q1 2020, based on a request for proposals which was issued to several database providers. The database for the WFH GTR will begin development in Q2 2020, with the aim of having a final database ready for launch in by end of 2020, when the first gene therapy product is available to patients. At this time, we will also begin recruitment of patients who have received gene therapy through a clinical trial.

Patients will be recruited through hemophilia treatment centers (HTC) who provide gene therapy to patients with hemophilia. Investigators will recruit patients into the WFH GTR and enter baseline and follow up data over the long term. There is no determined end date for this registry. For countries who have an existing national registry, we offer the possibility of linking databases directly.

ELIGIBILITY:
Inclusion Criteria:

* People with hemophilia who have received a gene therapy product

Exclusion Criteria:

* None

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All people with hemophilia who have received a gene therapy product
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2050-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in long term safety: adverse events of interest | From baseline, through study completion (15 years)
  Months 3, 6, 9, 12, 18, 24; and annually thereafter for 15 years.
Change in efficacy: factor level and bleeding events | From baseline, through study completion (15 years)
  Months 3, 6, 9, 12, 18, 24; and annually thereafter for 15 years.